CLINICAL TRIAL: NCT01258257
Title: EARLYdrain - Prospective Outcome Study of Early Lumbar Drainage in Aneurysmal Subarachnoid Hemorrhage
Brief Title: EARLYdrain - Outcome After Early Lumbar CSF-drainage in Aneurysmal SAH
Acronym: EARLYDRAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Stefan Wolf, Stefan Wolf, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EARLYDRAIN
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Aneurysm; Subarachnoid hemorrhage; Lumbar drain; Cerebral vasospasm; Cerebral Ventricles; Cerebrospinal Fluid; Prospective Studies; Drainage/methods*; Humans; Subarachnoid Hemorrhage/cerebrospinal fluid*; Subarachnoid Hemorrhage/complications*; Subarachnoid Space/surgery*; Vasospasm, Intracranial/etiology; Vasospasm, Intracranial/surgery*
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Vasospasm, Intracranial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbar drain (LD) / Tuohy drain (Active Comparator): Intervention: Insertion of a lumbar drain All patients in the LD group receives a lumbar drain during anesthesia required for aneurysm treatment. Drainage of CSF is started after the post-procedural CT scan on day one after aneurysm securement.
  Interventions: Procedure: Insertion of a lumbar drain
- No Lumbar drain (NoLD) (No Intervention): Patients randomized to the control group should not receive a lumbar drain before the planned control angiography to be performed on day 7 to 10 after SAH. If the patient develops hydrocephalus, and no EVD was placed initially for CSF drainage, a lumbar drain may be installed at the discretion of the local investigator. These patients are analyzed in the intention-to-treat analysis, but are not suitable for per-protocol analysis.

INTERVENTIONS:
Procedure: Insertion of a lumbar drain — In patients in the LD group, after insertion of the drain CSF is drained slowly and steadily at a rate of approximately 5 ml per hour. This leads to a planned daily CSF drainage of about 120 ml per day via lumbar route. To facilitate accuracy of drainage, regular drainage control every other hour and stopping in case of unwarranted excess drainage is strongly recommended by the principal investigators. In case of neurological decline suspiciously related to the lumbar drainage, the drain is closed immediately and may be gradually restarted after 12 to 24 hours, after performing a CCT scan. The drain is planned to remain in place until the control angiography on day 7 to 10 after the initial hemorrhage.
  Other Names: Tuohy drain
  Arms: Lumbar drain (LD) / Tuohy drain

SUMMARY:
The intention of the study is to investigate whether drainage of cerebral spinal fluid via a lumbar route ("Tuohy-drain") will improve outcome after intracranial aneurysmal subarachnoid hemorrhage (SAH).

DETAILED DESCRIPTION:
1. Introduction

   Patients suffering from aneurysmal subarachnoid hemorrhage (SAH) are predominantly threatened by two distinct medical problems. Firstly, they may experience a second - and often more severe - hemorrhage, and secondly, they may suffer a constringence reaction of the vessels supplying the brain with blood, called vasospasm.

   The first problem is resolved by rapid cerebrovascular imaging and subsequent treatment of the ruptured aneurysm, thus preventing recurrent hemorrhage. Aneurysm treatment may be performed either via craniotomy and surgical clipping of the aneurysm or with endovascular techniques by occluding the aneurysm with small platinum coils.

   The vasospasm - the second problem - is more difficult to handle. A hypothesis is that the development of vasospasm is related to the amount of blood in the basal cisterns. Therefore, a possible strategy tries to remove this blood as much as possible. Excess removal of cerebral spinal fluid (CSF) via an external ventricular drain fails in preventing vasospasm and may lead to a higher incidence of posthemorrhagic shunt dependency. Reason is that after aneurysmal SAH, the blood is packed more densely in the basal cisterns and therefore only CSF, being more lightweight, is drained from the ventricles. As an alternative approach, application of a lumbar drain is proposed to address clotting of the blood in the basal cisterns. Three retrospective studies in patients after aneurysmal SAH, the newest being available only as abstract, were able to establish the safety of this approach (Klimo et al, Kwon et al, Tizi et al (abstract DGNC 2009)). One of the fully published studies addressed vasospasm prophylaxis after surgical clipping, while the other was performed in patients after endovascular coiling. All studies led to a markedly diminished incidence of angiographic vasospasm. Therefore, a prospective study addressing the efficacy of this novel therapeutic approach is warranted.

   The focus of the EARLYDRAIN study is to examine the efficacy of application of lumbar drainage in patients with acute subarachnoidal hemorrhage from a cerebral aneurysm. Hypothesis is that early application of lumbar drainage after aneurysmal SAH leads to a diminished incidence of cerebral vasospasm, as assessed by digital subtraction angiography, and an improved outcome, measured by the modified Rankin score, at six months.
2. Study outline

   Patients suffering from aneurysmal SAH are treated according to international standards. Aneurysm treatment is at the discretion of the neurovascular team taking care for a patient and not specified by the study protocol. All medical treatment is performed according to local guidelines and standard operating procedures.

   Any patient meeting the inclusion criteria and not violating the exclusion criteria may participate in the EARLYDRAIN study and be randomized to either receive a lumbar drain or not, thus defining the two distinct groups LD and NoLD. To prevent premature rupture of the aneurysm due to accidental drainage, randomization to the study and eventual placement of a lumbar drain takes place after securing the aneurysm by the preferred method of choice. Any patient in the LD group receives a lumbar drain during anesthesia required for aneurysm treatment. This is to be performed before anticoagulation or anti-platelet therapy is initiated, which sometimes is warranted after endovascular coiling. A post-procedural CCT scan of the brain is performed within to 24 hours of aneurysm treatment. In case of any neurological worsening after the procedure it is strongly recommended to perform the follow-up CCT scan as soon as possible.

   In patients in the LD group, CSF drainage is started via LD slowly and steadily at a rate of approximately 5 ml per hour after the post-interventional CCT. This leads to a planned daily CSF drainage of about 120 ml per day via lumbar route. Patients in both groups may receive additional CSF drainage via a ventricular device as required. The amount of CSF drained via ventricular route is according to clinical requirement and not specified.

   To facilitate accuracy of drainage, regular drainage control every other hour and stopping in case of excess drainage is strongly recommended by the principal investigators. In case of neurological decline suspiciously related to the lumbar drainage, the drain is closed immediately and may be gradually restarted after 12 to 24 hours, after performing a CCT scan.

   If the post-procedural CCT or any other follow-up CCT scan shows absent basal cisterns or any signs of threatening herniation, lumbar CSF diversion in the LD group shall not be performed. It may still be feasible to carefully drain CSF via the lumbar route may (Tuettenberg et al), but this is at the discretion of the local investigator and not recommended.

   In patients requiring sedation and mechanical ventilation, either due to neurological impairment or otherwise, intracranial pressure monitoring is mandatory. This may be performed according to local policy either with parenchymal or ventricular devices. If the intracranial pressure exceeds 20 mmHg, further CSF drainage via lumbar route shall be interrupted until the ICP is below 20 mmHg again. Careful CSF drainage via the lumbar route may be still feasible in case of high intracranial pressure (Tuettenberg et al), but is at the discretion of the local investigator.

   Further neuromonitoring with TCD, EEG, brain tissue oxygenation, jugular bulb oxymetry, regional cerebral blood flow, microdialysis or other devices is at the discretion of the center and according to its local guidelines. As far as possible, this data should be saved electronically for post-hoc analysis.

   A CCT scan as well as conventional digital subtraction angiography, CT angiography or MR angiography for assessment of vasospasm in the larger vessels is routinely performed on day 7 to 10 after the initial hemorrhage, regardless of the patient condition. In case of clinical suspicion of vasospasm, angiography may be performed at any time. If it is performed earlier and the patient shows no clinical deterioration thereafter, the angiography on day 7 to 10 is omitted.

   After cerebrovascular imaging on day 7 to 10, or day 8 in case of an earlier angiography, the lumbar drainage of CSF is stopped in the LD group. It may be pursued on a clinical base, as required.

   Amount and duration of CSF drainage Patients randomized to the lumbar drainage group shall receive a daily drainage of 120 ml CSF, or 5 ml per hour for seven days. If higher amounts of CSF need to be drained on clinical grounds as in patients with hydrocephalus, this is preferably performed via external ventricular drain.

   The drain is planned to remain in place until the control angiography on day 7 to 10 after the initial hemorrhage. The local investigator may decide to remove the drain earlier in patients fully mobilized without clinical necessity of CSF drainage. However, consecutive drainage should not be less than four days to achieve a valid study result. Lumbar CSF drainage may be prolonged beyond the control angiography on clinical requirement. The amount of CSF drainage may then be adjusted to clinical needs and bears no further restriction.

   Patients randomized to the control group should not receive a lumbar drain before the planned control angiography to be performed on day 7 to 10 after SAH. If the patient develops hydrocephalus, and no EVD was placed initially for CSF drainage, a lumbar drain may be installed at the discretion of the local investigator. These patients are analyzed in the intention-to-treat analysis, but are not suitable for per-protocol analysis.
3. Consent to the study

   Consent for study inclusion is sought after explanation and agreement to a specific aneurysm treatment. Thus, patients capable of consenting to the aneurysm treatment get the study details explained themselves and may or may not agree to participate. If a patient is incapable for consenting to the proposed treatment, the legal representative should be informed on the conditions of treatment choices and afterwards, on the details of the EARLYDRAIN study. A patient may be randomized if the legal representative gives informed consent to the study, based on the presumed will of the patient. If neither the patient is capable of giving informed consent nor a legal representative is available in due time, an independent physician not involved in the patient's treatment nor in the trial may be asked for study approval. In these cases of deferred consent, a legal representative needs to be established as soon as possible, according to German law. As soon as a legal representative is available and/or the patient is capable again to consent to the study, he or she must be asked to give informed consent. If the patient or his/her legal representative refuses consent after inclusion by advice of an independent physician, no further study participation of the patient is possible. In this case, however, the patient or his/her legal representative are asked to give consent for evaluation of already acquired data.
4. Safety of lumbar drains after aneurysmal SAH

   In all three retrospective studies, mortality was lower in the lumbar drainage group. None of the retrospective studies mentions procedural related complications for the lumbar drains (Klimo et al, Kwon et al, Tizi et al (abstract at the DGNC 2009)). In patients with increased intracranial pressure, careful lumbar drainage of CSF may be a possible treatment even in case of compressed basal cisterns (Tuettenberg et al). To date, there is no data available indicating an increased risk of lumbar drainage in a controlled neurointensive care environment.
5. Insurance coverage

As the EARLYDRAIN study compares two standard procedures of CSF drainage after subarachnoid hemorrhage used in clinical routine, no additional patient insurance is necessary to perform the study. German laws §§ 40 to 42 Arzneimittelgesetz or §§ 20 to 23 Medizinproduktegesetz are not applicable. Any hypothetical adverse events of either treatment are covered by the regular treatment contracts which do include clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* First aneurysmal SAH
* Pre-morbid modified Rankin Scale score 0 or 1
* Aneurysm treatment performed in the first 48 hours after the initial hemorrhage.
* Informed consent by the patient or his/her legal representative. In case neither the patient is capable of giving informed consent nor a legal representative is available, informed consent can be given by an independent physician neither involved in the patient´s treatment nor the trial (for specification see below)

Exclusion Criteria:

* Subarachnoid hemorrhage of other than aneurysmal origin
* No hemorrhage visible on initial CCT scan (Fisher Grade I)
* Pregnancy
* Concurrent participation in another interventional trial (participation in an observational trial is allowed)
* Life expectancy less than 1 year for other reasons than the actual SAH
* Other concomitant severe disease that would confound with treatment
* Other clear contraindication for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Disability in Lumbar drainage group (LD) vs. disability in control group (No-LD) | 6 months after SAH
  Disability is assessed by the modified Rankin Scale, dichotomized at a score of 0 to 2 versus 3 to 6 (6=death).Assessment is performed by a blinded investigator of the local study center by personal visit. Alternatively, a telephone questionnaire is suitable for outcome assessment of the modified Rankin Scale (13). Outcome assessment is planned to be done on the whole dataset as well as in preplanned stratified subsets (i.e. for example clinical SAH grade according to the Hunt&Hess scale 1-2 vs. 3-5 (14), CT grading according to Fisher I-III vs. IV (15)).

SECONDARY OUTCOMES:
mortality | 6 months after SAH
Modified Rankin scale (mRS) score as continuous variable | 6 months after SAH
Angiographically determined vasospasm | once between day 7 to 9 after SAH
  Vasospasm here is defined as a caliber reduction by 33% or more on day 7-9 compared to the initial digital subtraction angiography.
Vasospastic infarction | last CT-scan during hospital stay, an expected average of 4 weeks
Expression of clinical delayed neurological deficit | day 1-14 after SAH
Transcranial duplex ultrasound measured flow velocity in both middle cerebral arteries | daily during hospital stay of the patient
  TCD-measured mean flow velocity in both MCA is determined daily at a depth of 50-60 mm.
Early mortality | Time span of initial hospital treatment after SAH, an expected average of 4 weeks
Rate of CSF shunt insertion in the first six months | First 6 months after SAH
Presence of CSF infection | First 14 days after SAH
  Infection in this case is defined by the modified criteria for device-associated (CDC) meningitis (treatment required on either positive culture, or elevated cell count, red cell/ white cell ratio, increased lactate and/or decreased glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Wolf, Dr., Principal Investigator — Charite University medicine / department of neurosurgery
Locations (1):
- Charité University Medicine Department of Neurosurgery Campus Virchow Klinikum, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Full anonymized data is planned to be shared among collaborators.

REFERENCES:
- [Background] Klimo P Jr, Kestle JR, MacDonald JD, Schmidt RH. Marked reduction of cerebral vasospasm with lumbar drainage of cerebrospinal fluid after subarachnoid hemorrhage. J Neurosurg. 2004 Feb;100(2):215-24. doi: 10.3171/jns.2004.100.2.0215. PMID 15086227
- [Background] Kwon OY, Kim YJ, Kim YJ, Cho CS, Lee SK, Cho MK. The Utility and Benefits of External Lumbar CSF Drainage after Endovascular Coiling on Aneurysmal Subarachnoid Hemorrhage. J Korean Neurosurg Soc. 2008 Jun;43(6):281-7. doi: 10.3340/jkns.2008.43.6.281. Epub 2008 Jun 20. PMID 19096633
- [Background] Tuettenberg J, Czabanka M, Horn P, Woitzik J, Barth M, Thome C, Vajkoczy P, Schmiedek P, Muench E. Clinical evaluation of the safety and efficacy of lumbar cerebrospinal fluid drainage for the treatment of refractory increased intracranial pressure. J Neurosurg. 2009 Jun;110(6):1200-8. doi: 10.3171/2008.10.JNS08293. PMID 19249925
- [Derived] Truckenmueller P, Wolf S, Wasilewski D, Vajkoczy P, Fruh A; Earlydrain Study Group. Association of Fluid Balance and Hemoglobin Decline With Neurological Outcome After Aneurysmal Subarachnoid Hemorrhage. Crit Care Med. 2024 Sep 1;52(9):1391-1401. doi: 10.1097/CCM.0000000000006332. Epub 2024 May 21. PMID 38775857
- [Derived] Fruh A, Truckenmuller P, Wasilewski D, Vajkoczy P, Wolf S; Earlydrain Study Group. Analysis of Cerebral Spinal Fluid Drainage and Intracranial Pressure Peaks in Patients with Subarachnoid Hemorrhage. Neurocrit Care. 2024 Oct;41(2):619-631. doi: 10.1007/s12028-024-01981-9. Epub 2024 Apr 15. PMID 38622488
- [Derived] Wolf S, Mielke D, Barner C, Malinova V, Kerz T, Wostrack M, Czorlich P, Salih F, Engel DC, Ehlert A, Staykov D, Alturki AY, Sure U, Bardutzky J, Schroeder HWS, Schurer L, Beck J, Juratli TA, Fritsch M, Lemcke J, Pohrt A, Meyer B, Schwab S, Rohde V, Vajkoczy P; EARLYDRAIN Study Group. Effectiveness of Lumbar Cerebrospinal Fluid Drain Among Patients With Aneurysmal Subarachnoid Hemorrhage: A Randomized Clinical Trial. JAMA Neurol. 2023 Aug 1;80(8):833-842. doi: 10.1001/jamaneurol.2023.1792. PMID 37330974
- [Derived] Bardutzky J, Witsch J, Juttler E, Schwab S, Vajkoczy P, Wolf S. EARLYDRAIN- outcome after early lumbar CSF-drainage in aneurysmal subarachnoid hemorrhage: study protocol for a randomized controlled trial. Trials. 2011 Sep 14;12:203. doi: 10.1186/1745-6215-12-203. PMID 21917146